CLINICAL TRIAL: NCT01039545
Title: Symptomatic Therapy of Uncomplicated Lower Urinary Tract Infections in the Ambulatory Setting. A Randomized, Double Blind Trial
Brief Title: Symptomatic Therapy of Uncomplicated Lower Urinary Tract Infections in the Ambulatory Setting.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: New power calculation (reduction of necessary patient number)
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Clinic for Infectious Diseases, University Hospital Bern, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 254/09
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Urinary Tract Infections
Keywords: Urinary tract infections; Anti-bacterial agents
MeSH Terms: conditions — Urinary Tract Infections | interventions — Diclofenac; Norfloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- antibiotic (Active Comparator): Norfloxacin for three days, followed by fosfomycin on day 4 if deemed necessary
  Interventions: Drug: Norfloxacin
- symptomatic (Experimental): Diclofenac retard for three days, followed by fosfomycin on day 4 if deemed necessary
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac — Diclofenac retard 75mg twice daily for 3 days, followed by fosfomycin 3g single dose on day 4 if deemed necessary
  Arms: symptomatic
Drug: Norfloxacin — Norfloxacin 400mg twice daily for 3 days, followed by fosfomycin 3g single dose on day 4 if deemed necessary
  Arms: antibiotic

SUMMARY:
We propose to perform a randomized controlled patient and assessor blind trial in women between the ages of 18 to 70 years with acute uncomplicated UTI to evaluate initial symptomatic treatment for 3 days with the non-steroidal anti-inflammatory drug diclofenac (experimental intervention) against immediate antibiotic treatment with norfloxacin for 3 days (control intervention). Both interventions are followed by optional delayed antibiotic treatment with single dose fosfomycin if deemed necessary by the patients. The primary objective is to determine whether initial symptomatic treatment followed by optional delayed antibiotic treatment (experimental intervention) is non-inferior to immediate antibiotic treatment (control intervention) in terms of symptom resolution.

DETAILED DESCRIPTION:
Background

Urinary tract infection (UTI) is the most frequent bacterial infection diagnosed and treated by general practitioners and accounts for about 15% of antibiotic prescriptions in ambulatory medicine. World-wide raise of antibiotic resistance among uropathogens, most commonly Escherichia coli, threatens treatment of UTI. Uncomplicated UTI, the most frequent manifestation of UTI, is a benign, self-limited disease and the primary goal of treatment is symptom relief not cure. Antibiotic treatment reduces the duration of symptoms by 1-2 days from 5-6 days to 3-4 days. Symptoms of cystitis are the result of an inflammation evoked by bacterial products which stimulate the production of prostaglandins by a cyclooxygenase dependent mechanism. Therefore, we propose that symptom control with a non-steroidal anti-inflammatory drug (NSAID), an inhibitor of cyclooxygenase 1 and 2, may be equally effective for symptom control as standard antibiotic therapy in non-complicated UTI and may therefore help to reduce antibiotic consumption.

Objective

The primary objective is to determine whether initial symptomatic treatment followed by optional delayed antibiotic treatment (experimental intervention) is non-inferior to immediate antibiotic treatment followed by optional delayed antibiotic treatment (control intervention) in terms of symptom resolution.

The secondary objective is to determine whether the experimental intervention is superior to control in reducing the proportion of patients undergoing antibiotic treatment.

Methods

Randomized controlled patient and assessor blind trial performed in general practices. Study population are women between the ages of 18 to 70 years with acute uncomplicated UTI. The experimental intervention will consist of symptomatic treatment with diclofenac 75mg twice daily, followed by optional, delayed antibiotic treatment with single dose of 3g fosfomycin if deemed necessary by the patient. The control intervention will consist of immediate antibiotic treatment with norfloxacin 400mg twice daily for three days, followed by optional, delayed antibiotic treatment with single dose of 3g fosfomycin if deemed necessary by the patient. Patients will use a diary to describe symptoms for 10 days. A follow-up telephone interview will be performed on day 10 and 30.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age between 18 and 70 years
* Written informed consent
* At least one typical symptom of acute, lower urinary tract infection out of dysuria, frequency, macrohaematuria, cloudy or smelly urine or self-diagnosed cystitis
* A urine dipstick test should be indicative of UTI by positive nitrite or leucocyturia

Exclusion Criteria

* Duration of UTI symptoms for more than 7 days before physician's visit
* Clinical signs of invasiveness such as fever (axillary body temperature >38 degrees Celsius), costovertebral pain or tenderness, rigors, nausea or vomiting
* Known or suspicion of anatomical or functional abnormality of the urinary tract
* Vaginal symptoms: discharge, irritation
* Diabetes mellitus
* Immunosuppression (e.g. prednisone equivalent >10mg per day for >14 days, chemotherapy, radiotherapy, immunomodulators, HIV infection, neutropenia)
* Any other serious comorbidity as judged by the treating physician
* Bladder catheter in situ or during the past 30 days
* Pregnancy
* Recurrent urinary tract infection (more than 3 infections during the last 12 months)
* Antibiotic treatment during the last 4 weeks
* Hypersensitivity to one of the study medications
* Psychiatric illness or dementia
* Unable to communicate in German or French language
* Documented coagulopathy (including therapy with coumarine derivatives) or documented history of gastric or duodenal ulcer disease
* Documented renal insufficiency grade III or higher (calculated GFR <60) or known congestive heart failure (NYHA III or higher)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with resolution of symptoms on day 4 | one month

SECONDARY OUTCOMES:
The proportion of patients ever on antibiotics between randomization at day 1 and follow-up at day 30 | one month
The proportion of patients using single dose fosfomycin on day 4 | one month
The proportion of patients with re-consultations because of UTI within 30 days | one month
The mean composite symptom scores on days 4, 7 and 30 | one month
The proportion of patients with resolution of symptoms on day 7 | one month
The proportion of patients with complete resolution of symptoms on days 4 and 7 | one month
The time until resolution of symptoms | one month
The proportion of patients with adverse events | one month
Mean overall patient stratification | one month
Health-related quality of life on day 4 | one month
Number of working days lost | one month

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kronenberg, Principal Investigator — University of Bern
Locations (1):
- Institute for Infectious Diseases, University of Berne, Bern, Switzerland

REFERENCES:
- [Derived] Sachdeva A, Rai BP, Veeratterapillay R, Harding C, Nambiar A. Non-steroidal anti-inflammatory drugs for treating symptomatic uncomplicated urinary tract infections in non-pregnant adult women. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD014762. doi: 10.1002/14651858.CD014762.pub2. PMID 39698942
- [Derived] Kronenberg A, Butikofer L, Odutayo A, Muhlemann K, da Costa BR, Battaglia M, Meli DN, Frey P, Limacher A, Reichenbach S, Juni P. Symptomatic treatment of uncomplicated lower urinary tract infections in the ambulatory setting: randomised, double blind trial. BMJ. 2017 Nov 7;359:j4784. doi: 10.1136/bmj.j4784. PMID 29113968